CLINICAL TRIAL: NCT00541905
Title: Prospective, Single-arm, Multicenter Trial to Investigate the Efficacy and Safety of NT 201 and the Duration of Treatment Effect After One Injection Session and in Long-term Treatment in Patients With Cervical Dystonia
Brief Title: Daily Dystonia Practice - A Trial to Investigate NT 201, the Duration of Treatment Effect After One Injection Session and in Long-term Treatment in Cervical Dystonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRZ 60201-0605/1; 2006-003410-18 (EudraCT Number)
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — incobotulinumtoxinA

ARMS (1):
- NT 201 (50-300 Units) (Experimental): NT 201 (Xeomin®, also know as IncobotulinumtoxinA or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection.
  Interventions: Drug: NT 201

INTERVENTIONS:
Drug: NT 201 — Subjects to receive up to 5 injection sessions, with a total dose of up to 300 Units each. No more than 50 units should have be given at any one injection site during one session.

SUMMARY:
The aim of this study is to confirm efficacy and safety of NT 201 (Xeomin®, also known as IncobotulinumtoxinA) after one injection session and to determine the efficacy and safety profile and the duration of treatment effect of NT 201 in long-term treatment with repeated injection sessions.

ELIGIBILITY:
Inclusion Criteria:

* Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) - total score at baseline > / = 25 with TWSTRS - severity score > / = 10 and TWSTRS - disability score > / = 3
* Patients must be on a stable dose of other medications
* For pre-treated patients only: Source documentation of the last two consecutive injection sessions with botulinum neurotoxin type A and stable treatment response directly prior to trial entry
* For pre-treated patients only: At least 10 weeks must have passed between the last injection session of botulinum neurotoxin type A for cervical dystonia and the time of the baseline visit.
* For pre-treated patients only: The most recent injection session with botulinum neurotoxin for cervical dystonia must have been at a dose of ≤ 300 units of Botox® or Xeomin®, or ≤ 1,200 units Dysport®.
* Age > / = 18 and < 76 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS), total score: Change from study baseline (initial injection session) to week 4 | From baseline to week 4

SECONDARY OUTCOMES:
TWSTRS, Single interventional effect | From week 10-24 to week 14-28, from week 20-48 to week 24-52, from week 30-72 to week 34-76, and from week 40-96 to week 44-100
  Single interventional effect of one injection session by the change of the TWSTRS total, severity and disability scores from each cycle baseline to 4 weeks thereafter.
TWSTRS, overall interventional effect | From study baseline to week 14-28, 24-52, 34-76, and 44-100
  Measured by the change in the TWSTRS total, severity and disability scores, from study baseline to each examination 4 weeks after the injection sessions
Global Assessment of Efficacy by Investigator (GAEI) | Week 10-24, 20-48, 30-72, and 40-96
  At the end of each injection cycle
Subject Evaluation of Global Response (PEGR) | Week 10-24, 20-48, 30-72, and 40-96
  At the end of each injection cycle.
Time from last injection session to onset of treatment effect as given by subjective subject assessment | Up to 4 weeks from last injection session
  Measured in days.
Time from last injection session to waning of treatment effect as rated by subjective subject assessment | Up to 24 weeks from last injection session
  Measured in weeks.
Duration of treatment effect | Up to 24 weeks from last injection session
  Defined as time period within an injection cycle from the day of the injection session until the day where the need for reinjection was indicated by the subject (if subject experienced an onset of treatment effect).
Dystonia Discomfort Scale (DDS) score (subject diary), change from baseline | From study baseline up to week 100

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dirk Dressler, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Medizinische Hochschule Hannover (LKP), Hanover, Germany

REFERENCES:
- [Result] Dressler D, Kupsch A, Paus S, Seitzinger A, Gebhardt B. Sustained efficacy of Incobotulinumtoxin-A (Xeomin®; Botulinum Neurotoxin Type-A, free from Complexing Proteins) in Long-Term Treatment of Cervical Dystonia. European Journal of Neurology 18 (Suppl. 2): 482, 2011.
- [Result] Dressler D, Paus S, Seitzinger A, Gebhardt B, Kupsch A. Long-term efficacy and safety of incobotulinumtoxinA injections in patients with cervical dystonia. J Neurol Neurosurg Psychiatry. 2013 Sep;84(9):1014-9. doi: 10.1136/jnnp-2012-303608. Epub 2013 May 18. PMID 23687362